CLINICAL TRIAL: NCT06087939
Title: Outcome and Predictors of Mortality of Patients on Prolonged Mechanical Ventilation in Critically Ill Patients: a Multicenter Retrospective Cohort Study
Brief Title: Outcome and Predictors of Mortality of Patients on Prolonged Mechanical Ventilation
Status: Not yet recruiting | Type: Observational
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Sara Timerga, Lecturer, Wollo University
Other Study IDs: PMV
Record Dates: First submitted 2023-09-29; First posted 2023-10-18 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Outcome
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical ventilation — Mechanical ventilation (MV) is a life support technique that is routinely used in the intensive care units (ICUs) for patients with life-threatening conditions.

SUMMARY:
Prolonged mechanical ventilation (PMV) and weaning failure are factors associated with prolonged hospital length of stay and increased morbidity and mortality. In addition to the individual challenges that stress patients and their families, the resource-intensive care these patients receive places a significant burden on the public health system. These burdens often persist over the long term, especially in the case of weaning failure with subsequent home mechanical ventilation (HMV).

This study will provide invaluable and in-depth knowledge of major sources of admission to ICU and will clarify the cause for the outcomes seen after prolonged mechanical ventilation in ICU admission, at Dessie comprehensive Hospital, the result of our study will also serve as a source or baseline information for future valuable researches to be undergone around the subject of interest.

DETAILED DESCRIPTION:
The number of patients requiring prolonged mechanical ventilation after acute illness is increasing. Their long-term outcome is poor and has not improved significantly over the past 20 years. The symptom burden for patients is considerable, and family members often suffer from significant physical and emotional strain. Long-term survivors report lasting physical limitations, but their emotional health is generally good. Care for many patients requiring prolonged mechanical ventilation is shifting t post-intensive care unit settings. While this trend has resulted in cost savings for hospitals and payers, it has not had a major impact on patient outcomes.

Patients requiring prolonged mechanical ventilation consume a disproportionate amount of healthcare resources and clinician time. Measurement and knowledge of their outcomes will guide efforts to improve their care.

This study will be conducted in Dessie Comprehensive Specialized Hospital from August 2023 to January 2024. A retrospective cohort study will be conducted. Data will be checked, coded, entered, and analyzed using SPSS version 22 software. Descriptive statistics will be used to summarize data, tables, and figures for display results. Bivariate and multivariate analyses will be used to see the effect of the independent variable on the outcome variable. Variables that are significant on bivariate analysis at a p-value less than 0.2 will be taken to multivariate analysis. In multivariate analysis, a p-value of less than 0.05 will be used as a cut-off point for the presence of association. The strength of the association will be measured by 95% confidence interval and odd ratio.

ELIGIBILITY:
Inclusion Criteria:

* All charts of critically ill patients on prolonged mechanical ventilation in of Dessie Comprehensive Specialized Hospital during the study period.

Exclusion Criteria:

* Charts with incomplete information and missing values as well as those that are not available will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All charts of critically ill patients admitted to ICU of Dessie comprehensive specialized hospital.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
clinical outcomes of critically ill patients undergoing prolonged mechanical ventilation | 5 months
  Clinical outcome: indicated either patient survived or died at the time of discharge.
  Prolonged mechanical ventilation: is defined as successful extubation after more than three spontaneous breathing trials or taking more than 14 days

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the individual participant data when asked.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with 5 month time.